CLINICAL TRIAL: NCT03896568
Title: Phase I Clinical Trial of Allogeneic Bone Marrow Human Mesenchymal Stem Cells Loaded With A Tumor Selective Oncolytic Adenovirus, DNX-2401, Administered Via Intra-Arterial Injection in Patients With Recurrent High-Grade Glioma
Brief Title: MSC-DNX-2401 in Treating Patients With Recurrent High-Grade Glioma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: DNAtrix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0953; NCI-2019-01195 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0953 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: IDH1 wt Allele; Recurrent Anaplastic Astrocytoma; Recurrent Glioblastoma; Recurrent Gliosarcoma; Recurrent Malignant Glioma
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Gliosarcoma; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part I (oncolytic adenovirus Ad5-DNX-2401) (Experimental): Patients receive oncolytic adenovirus Ad5-DNX-2401 IA over 20-30 minutes on day 0.
  Interventions: Biological: Oncolytic Adenovirus Ad5-DNX-2401
- Part II (oncolytic adenovirus Ad5-DNX-2401, surgery) (Experimental): Patients receive oncolytic adenovirus Ad5-DNX-2401 as in part I. After 2 weeks, patients undergo surgery, then receive oncolytic adenovirus Ad5-DNX-2401 IA over 20-30 minutes.
  Interventions: Biological: Oncolytic Adenovirus Ad5-DNX-2401; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Biological: Oncolytic Adenovirus Ad5-DNX-2401 — Given IA
  Other Names: Ad5-Delta24RGD; DNX-2401; DNX2401; Oncolytic Ad5-Delta 24RGD; Oncolytic Adenovirus Ad5-Delta 24RGD
Procedure: Therapeutic Conventional Surgery — Undergo surgery
  Arms: Part II (oncolytic adenovirus Ad5-DNX-2401, surgery)

SUMMARY:
This phase I trial studies best dose and side effects of oncolytic adenovirus DNX-2401 in treating patients with high-grade glioma that has come back (recurrent). Oncolytic adenovirus DNX-2401 is made from the common cold virus that has been changed in the laboratory to make it less likely to cause an infection (such as a cold). The virus is also changed to target brain cancer cells and attack them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximal tolerated dose (MTD) of allogeneic bone marrow-derived human mesenchymal stem cells (BM-hMSCs) loaded with the oncolytic adenovirus DNX-2401 (BM-hMSCs-DNX2401) administered by intra-arterial injection (i.e., transfemoral endovascular intracranial injection) in patients with recurrent glioblastoma (GBM), IDH-mutant astrocytoma grade 4, gliosarcoma, or wild-type IDH-1 anaplastic astrocytoma.

II. To determine the local and systemic toxicity of allogeneic BM-hMSCs-DNX2401 administered by intra-arterial injection (i.e., transfemoral endovascular intracranial injection) in patients with recurrent GBM, gliosarcoma or wild-type IDH-1 anaplastic astrocytoma.

III. To determine at the molecular and cellular level the capacity of allogeneic BM-hMSCs-DNX2401 administered intra-arterially to home to and deliver DNX-2401 to recurrent GBM, gliosarcoma or wild-type IDH-1 anaplastic astrocytoma by analyzing post-treatment surgical brain tumor specimens for the expression and distribution of adenoviral proteins.

SECONDARY OBJECTIVES:

I. To assess shedding of adenovirus into the blood, sputum, and nasopharynx after intra-arterial administration of BM-hMSCs-DNX2401 in patients with recurrent GBM, gliosarcoma or wild-type IDH-1 anaplastic astrocytoma.

II. To assess the development of anti-adenovirus antibodies after intra-arterial administration of BM-hMSCs-DNX2401 in patients with recurrent GBM, gliosarcoma or wild-type IDH-1 anaplastic astrocytoma.

III. To evaluate immune-mediated cytokine responses after intra-arterial administration of BM-hMSCs-DNX2401 in patients with recurrent GBM, gliosarcoma or wild-type IDH-1 anaplastic astrocytoma.

IV. To assess anti-tumoral activity and to determine progression-free survival (PFS) and overall survival (OS) after intra-arterial administration of BM-hMSCs-DNX2401 in patients with recurrent GBM, gliosarcoma or wild-type IDH-1 anaplastic astrocytoma.

OUTLINE: This is a dose-escalation study.

PART I: Patients receive one or two infusions of BM-hMSCs-DNX-2401 intra-arterially (IA) over 20-30 minutes on day 0. Dose level 1-5 will receive 1 infusion. Dose level 6 will receive 2 infusions.

PART II: Patients receive one or two infusions BM-hMSCs-DNX-2401 IA, depending on the highest dose that was tolerated in Part 1. After 2 weeks, patients undergo surgery where the tumor is removed, then receive intramural injection of BM-hMSCs-DNX-2401 into the resection cavity.

After completion of study treatment, patients in both part I and II are followed up on days 1, 4, 7, and 14 of month 1,every 6 weeks for 6 months (4 visits), then every 8 weeks for 1 year (6 visits), then every 4 months for 1 year (3 visits), then every 6 months until the tumor grows back. Patients treated at Dose level 6 in Part 1 and Part 2 are also followed up on Day 12, then on Day 1, 4, and 7 after second infusion, then on Day 1, 7, and 14 post-craniotomy for Part 2, Dose Level 6, then ,every 6 weeks for 6 months (4 visits), then every 8 weeks for 1 year (6 visits), then every 4 months for 1 year (3 visits), then every 6 months until the tumor grows back.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following inclusion criteria to be eligible and enroll:

1. Subjects must be willing and able to provide informed consent, undergo and comply with all study assessments, and adhere to the protocol schedule.
2. Patients with recurrent malignant GBM or gliosarcoma will be eligible. Patients with recurrent anaplastic astrocytoma with wild-type IDH-1 gene will also be eligible if there is a significant enhancing mass on MRI (≥1.0 cm in diameter with upper limit of 5 cm maximal diameter) because their prognosis/behavior is similar to GBM. Subjects with an initial diagnosis of an IDH-mutant grade 2 or 3 astrocytoma are also eligible at recurrence if a biopsy at recurrence is determined to be IDH-mutant grade 4 astrocytoma, and there is a significant enhancing mass on MRI (≥1.0 cm in diameter with upper limit of 5 cm maximal diameter). A pathology report constitutes adequate documentation of histology for study inclusion.
3. Patients must show unequivocal evidence for tumor recurrence or progression by MRI scan after failing prior surgical resection, biopsy, chemotherapy or radiation. A baseline MRI must be performed within 24 days prior to registration. Biopsy is encouraged at the time of recurrence if it is unclear that there is recurrent tumor. However, biopsy is not required if the practicing physician thinks that there is adequate radiographic and clinical evidence for recurrence.
4. Male or female patients ≥ 18 years of age.
5. Patients must be able to undergo endovascular treatment based on Doppler studies showing ICA that is less than 50% occluded.
6. For patients undergoing resection for biological endpoints, tumors must be surgically resectable at the time of baseline evaluation and craniotomy for tumor resection is indicated as part of their standard medical care.
7. Tumors must be ≥1.0 cm in diameter with upper limit of 5 cm maximal diameter.
8. Patients must have a Karnofsky performance score ≥ 70.
9. Patients must have a life expectancy of at least 16 weeks.
10. Patients must have adequate bone marrow function (absolute granulocyte count > 1,500 and platelet count of > 75,000), adequate liver function (SGPT and SGOT and bilirubin < 2 times institutional normal ranges), and adequate renal function (creatinine < 2.0 times institutional normal) prior to starting therapy.
11. Prothrombin time/international normalized ratio (PT/INR) or partial thromboplastin time (PTT) ≤ 1.5x ULN.
12. Subjects who have received the following chemotherapies must have completed them within the following time periods prior to Baseline/Day 0 of hMSC-DNX2401 delivery with recovery from any drug-related toxic effects to Grade 1, or less, severity:

    * Four weeks from cytotoxic agents (3 weeks from procarbazine or Temozolomide, 2 weeks from vincristine)
    * 6 weeks from nitrosoureas (CCNU, BCNU)
    * Four weeks from any targeted investigational agent
    * One week from non-cytotoxic agents
13. This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender.
14. No exclusion to this study will be based on race. Minorities will actively be recruited to participate. The malignant glioma patient population treated at MDACC over the past year is as follows:

    * American Indian or Alaskan Native - 0
    * Asian or Pacific Islander - <2%
    * Black, not of Hispanic Origin - 3%
    * Hispanic - 6%
    * White, not of Hispanic Origin - 88%
    * Other or Unknown - 2%
    * Total - 100%
15. Patients must be 8 weeks from radiotherapy to minimize the potential for MRI changes related to radiation necrosis that might be misdiagnosed as progression of disease, or 4 weeks if a new lesion, relative to the pre-radiation MRI, develops that is outside the primary radiation field (beyond 80% isodose line). However, if a biopsy is undertaken prior to these times and this biopsy documents histological evidence for recurrent disease, then patients will be eligible regardless of the time after radiation.
16. Patients must be willing to forego other cytotoxic and non-cytotoxic drug or radiation therapy against the tumor while enrolled in the study.
17. Women of childbearing potential must have a negative urine or serum pregnancy test at screening.
18. Subjects and their partners must be willing to use effective birth control during the study and for up to 6 months following administration of hMSC-DNX2401. Birth control that is acceptable to use in this study:

    * Using twice the normal protection of birth control (i.e., double-barrier) by using a condom AND spermicidal jelly or foam, or a diaphragm AND spermicidal jelly or foam. A spermicidal jelly or foam must be used in addition to a barrier method (e.g., condom or diaphragm)
    * Birth control pills ("The Pill")
    * Depot or injectable birth control
    * IUD (Intrauterine Device)
    * Birth Control Patch (e.g., Othro Evra®)
    * NuvaRing®
    * Surgical sterilization (i.e., tubal ligation or hysterectomy for women or vasectomy for men)

Exclusion Criteria:

1. Histology other than GBM, gliosarcoma, IDH wild-type astrocytoma grade III or IDH-mutant astrocytoma grade 4.
2. Tumor foci detected below the tentorium or beyond the cranial vault.
3. Tumor within the posterior fossa.
4. Tumor with leptomeningeal spread.
5. Difficulty in obtaining vascular access for percutaneous procedure.
6. Ipsilateral carotid stenosis (>50%, by Doppler studies).
7. Thrombophilias or primary hematological diseases.
8. Transfusions or medications (G-CSF) to treat pancytopenia or other hematological conditions < 28 days prior to Baseline/Day 0/hMSC-DNX2401 administration.
9. Biologic/immunotherapy within 2 weeks of baseline.
10. Clinical or laboratory evidence of inflammatory and/or autoimmune disorders.
11. Any contraindication for undergoing MRI such as: individuals with pacemakers, epicardial pacer wires, infusion pumps, surgical and/or aneurysm clips, shrapnel, metal prosthesis, implants with potential magnetic properties, metallic bodies in the eyes, etc. In addition, subjects must present with tumor that is evaluable by MRI.
12. Pregnant or nursing females.
13. Evidence of active uncontrolled infection or unstable or severe intercurrent medical conditions. All subjects must be afebrile (i.e., <38.0° Celsius [C]).
14. Any medical condition that precludes surgery or endovascular treatment
15. Alcoholism (dependency), alcohol or substance abuse within twelve (12) months prior to screening that has caused health consequences.
16. Immunocompromised subjects or those with autoimmune conditions, active hepatitis (Liver function tests > 2x normal) or human immunodeficiency virus (HIV) seropositivity.
17. Evidence of bleeding diathesis or use of anticoagulant medication or any medication that may increase the risk of bleeding that cannot be stopped prior to surgery. If the medication can be discontinued prior to DNX-2401 injection then the subject may be eligible following consultation with the Study Chair. Low weight heparin and Lovenox (enoxaparin) administered on a temporary limited basis for post procedure DVT prophylaxis is permitted.
18. History or current diagnosis of any medical or psychological condition that in the Investigator's opinion might interfere with the subject's ability to participate or inability to obtain informed consent because of psychiatric or complicating medical problems.
19. Encephalitis, multiple sclerosis or other central nervous system (CNS) infection or primary CNS disease that would interfere with subject evaluation.
20. Subjects with known Li-Fraumini Syndrome or with a known germ line deficit in the retinoblastoma gene or its related pathways.
21. Subjects with significant systemic or major illnesses including but not limited to: congestive heart failure, ischemic heart disease, cerebrovascular disease (history of strokes or TIAs in large vessel or small vessel distribution), kidney disease or renal failure, active liver disease, organ transplantation, or significant psychiatric disorder.
22. Enrollment in a concomitant therapeutic clinical study.
23. Any condition that prevents compliance with the protocol or adherence to therapy.
24. For patients enrolled in the biological endpoint phase of the study, patients will be excluded if in the assessment of the surgeon, after resecting the tumor, there is high likelihood of injecting BM-hMSC-DNX2401 into the ventricles.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-02-12 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) | Up to 28 days
  The MTD will be defined as the dose below the dose that results in greater than or equal to one-third of the subjects exposed who experienced grade 3 or 4 (except hematological, grade 4 required) toxicity according to National Cancer Institute Common Toxicity Criteria that is deemed to be at least "probably related" to the study drug (i.e., dose-limiting toxicity [DLT]).
Incidence of adverse events (AEs) | Up to 1 year
  AEs will be summarized both overall and by dose group and tabulated by severity, relationship to BM-hMSCs-DNX 2401and causality. The number and percentage of subjects experiencing AEs will be tabulated by body system/preferred term both overall and by dose group. When an AE occurs more than once, the maximum severity and causality will be counted.

SECONDARY OUTCOMES:
Tumor response | Up to 1 year
  Will be based upon change in tumor size by serial magnetic resonance imaging scans post injection.
Time to progression | Up to 1 year
Virus replication in tumor | Up to 1 year
  Detection of replicating delta-24-RGD-4C in tumor tissue will be done by immunohistochemistry against E1A protein and hexon protein.
Virus shedding | Up to 1 year
  Polymerase chain reaction of serum, nasopharyngeal secretions, and urine will be performed.
Immunogenicity based on adenoviral (AdV) antibodies | Up to 1 year
  Enzyme-linked immunosorbent assay (ELISA) will be used to detect AdV antibodies in serum and virus assays to determine antibody titers (anti-AdV5 antibody immunofluorescence) will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick F Lang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Chen SR, Chen MM, Ene C, Lang FF, Kan P. Perfusion-guided endovascular super-selective intra-arterial infusion for treatment of malignant brain tumors. J Neurointerv Surg. 2022 Jun;14(6):533-538. doi: 10.1136/neurintsurg-2021-018190. Epub 2021 Nov 25. PMID 34824133
- See also: MD Anderson Cancer Center — http://www.mdanderson.org